CLINICAL TRIAL: NCT07234747
Title: Comparison of the Effects of Structured Core Stabilization Exercise Training and Exergaming-Based Core Stabilization Training in Children With Juvenile Idiopathic Arthritis
Brief Title: Structured vs. Exergaming-Based Core Stabilization in Children With Juvenile Idiopathic Arthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Collaborators: Çam Sakura Şehir Hastanesi (Unknown); Istanbul University (Other)
Responsible Party: Principal Investigator, Irem Donmez, Physiotherapist, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IremDIUC
Record Dates: First submitted 2025-09-23; First posted 2025-11-18 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-11

CONDITIONS: Juvenile Idiopathic Arthritis (JIA)
Keywords: core stabilization; juvenile idiopathic arthritis; exergaming
MeSH Terms: conditions — Arthritis, Juvenile

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Structured Core Stabilization Exercise Training (Experimental)
  Interventions: Other: Structured Core Stabilization Exercise Training
- Exergaming-Based Core Stabilization Training (Experimental)
  Interventions: Other: Exergaming-Based Core Stabilization Training

INTERVENTIONS:
Other: Structured Core Stabilization Exercise Training — This group is currently undergoing a structured core stabilization training program, consisting of supervised exercises conducted twice a week for 45 minutes per session over a 12-week period. The training is performed on a balance board to enhance postural control and trunk stability.
  The core-focused exercises include quadruped stabilization, extremity lifts in crawling position, planks, push-ups, mountain climbers, squats, single-leg squats, and lunges. These exercises are designed to strengthen deep trunk muscles and improve neuromuscular coordination, balance, and overall functional movement. Sessions are supervised by a physiotherapist to ensure correct execution and progression.
  Arms: Structured Core Stabilization Exercise Training
Other: Exergaming-Based Core Stabilization Training — This group is currently participating in an exergaming-based core stabilization training program using the SEG-BOARD device, developed under the TÜSEB B Project. The program is conducted twice a week for 45 minutes per session over a 12-week period. Although the SEG-BOARD is not specifically designed for core stabilization, it is a general-purpose exergaming exercise platform. In this study, it is utilized to support core-focused training through interactive visual and auditory feedback that promotes engagement and motor control.
  Participants perform exercises targeting core strength and stability, including quadruped-position stabilization, extremity lifts, planks, push-ups, mountain climbers, squats, single-leg squats, and lunges. These exercises are adapted into the exergaming format to enhance motivation and participation, while supporting improvements in trunk control and postural stability. All sessions are supervised by a physiotherapist.
  Arms: Exergaming-Based Core Stabilization Training

SUMMARY:
Juvenile Idiopathic Arthritis (JIA) is the most common inflammatory, autoimmune, and chronic rheumatic disease of childhood (1). In individuals diagnosed with JIA, increased inflammation leads to joint swelling, tenderness, restricted range of motion, and pain (2,3). Over time, these symptoms may result in impaired movement and proprioception, reduced muscle strength, and gait abnormalities (2,3).

Although ongoing medical treatment has been demonstrated to be highly effective in suppressing inflammation in children with rheumatic diseases, persistent pain despite treatment may limit mobility and contribute to the development of kinesiophobia. This condition may lead to the adoption of a sedentary lifestyle (4). A sedentary lifestyle may subsequently result in reduced functional capacity and physical fitness, increased risk of social isolation, and a decline in overall quality of life (5).

According to the literature, physical activity in children with rheumatologic diseases has been shown to reduce inflammation, increase muscle strength, improve functional capacity and mental health, reduce fatigue, and enhance quality of life (6,7). Non-pharmacological therapeutic exercise interventions have been found effective in alleviating chronic disease-related symptoms in children and in preventing secondary complications (8). The effectiveness of exercise therapy in children with JIA has been demonstrated in several studies, with commonly used programs including balance, proprioception, resistance, and range of motion exercises (9). However, only a limited number of studies have incorporated core-focused stabilization exercises into treatment protocols for children with JIA.

Although Core Stabilization Training (CST) initially gained popularity among athletes, it has since been integrated into rehabilitation programs and applied across various patient populations (10,11). CST is defined as the ability to control muscle activation in the lumbo-pelvic region, which is necessary for spinal stabilization and for transferring core strength from the trunk to the extremities. CST has been shown to positively affect standing, sitting, balance, postural stability, and gait (12).

A review of the literature confirms that Core Stabilization Training (CST) has beneficial effects on quality of life, pain, cardiorespiratory fitness, and functional ability (13). In studies involving children with Juvenile Idiopathic Arthritis (JIA), CST interventions were typically applied over a period of 12 weeks, with 2-3 sessions per week. The outcomes observed in this population were consistent with findings in the broader literature, supporting the effectiveness of CST in children with JIA (14).

Exergaming has emerged as an innovative approach to integrating physical activity into daily life (15). In the literature, exercise programs utilizing exergaming across various populations are frequently encountered. These studies have demonstrated multiple benefits of exergaming, including promoting physical activity, reducing perceived exertion, adapting physical activity to individual needs, and improving physical fitness (16). In children diagnosed with JIA, exergaming programs have shown improvements in physical performance and exercise skills, as well as significantly enhanced patient satisfaction (17). However, to date, no study has been identified in the literature that investigates the use of exergaming-based core stabilization training specifically in children with JIA.

The aim of the study is to compare the effects of an exergaming-based core stabilization training program and a structured core stabilization training program on physical fitness and functional capacity in children with Juvenile Idiopathic Arthritis (JIA). The study is designed as a randomized controlled trial. Children diagnosed with JIA will be included and randomly assigned to one of two groups. One group will receive structured core stabilization training, while the other will receive core stabilization training through exergaming. Both interventions will be administered over a 12-week period, with sessions held twice per week, each lasting 45 minutes.

To the best of available knowledge, this will be the first study to investigate the effectiveness of a core stabilization exercise program using exergaming in this population. This study is expected to contribute valuable insights to the literature on improving physical fitness and functional capacity in children with Juvenile Idiopathic Arthritis (JIA). Furthermore, it will provide the first clinical and scientific evidence regarding the innovative use of exergaming as a method for delivering core stabilization exercises.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 8 and 13
* Having been diagnosed with JIA at least 6 months prior
* Willingness to participate in the study

Exclusion Criteria:

* Having a balance problem due to vestibular or neurological conditions
* Having undergone surgery in the last 6 months that may interfere with exercise participation
* Inability to comply with the exercise program

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2025-11-10 (Estimated); Study Completion 2026-01-10 (Estimated)

PRIMARY OUTCOMES:
30-Second Sit-to-Stand Test (30STST) | Change from baseline and after the exercise program (12 weeks later).
  This test assesses lower limb muscle endurance and functional strength. Participants will be asked to sit and stand from a standard chair as many times as possible within 30 seconds. The total number of complete repetitions will be recorded.
6-Minute Walk Test (6MWT) | Change from Baseline and after the exercise program (12 weeks later).
  The 6MWT evaluates submaximal aerobic capacity and functional endurance. Participants will be instructed to walk continuously for 6 minutes down a 30-meter corridor. The total distance covered in meters will be recorded.
10-Step Stair Climb Test | Change from Baseline and after the exercise program (12 weeks later).
  This test measures functional lower extremity strength and mobility. Participants will be asked to ascend 10 stairs as quickly and safely as possible. The time to complete the stair climb will be measured in seconds using a stopwatch.

SECONDARY OUTCOMES:
FitnessGram Physical Activity Test Battery-Curl-up Test | Change from baseline and after the exercise program (12 weeks later).
  The participant will begin the test in the supine position, knees flexed approximately 140 degrees, feet flat on the floor, and legs slightly apart. The participant's arms will be parallel to the floor and torso. The palm will be positioned on the floor with the fingers stretched out. The purpose of this test is to do as many sit-ups as possible at a given speed. A maximum of 75 shuttles counts. The number of shuttles performed at the end of the test will be recorded. The curl-up test will be used to evaluate the abdominal muscle strength and endurance of children.
FitnessGram Physical Activity Test Battery-Push-up Test | Change from baseline and after the exercise program (12 weeks later).
  The participant will begin the test in the prone position, with their hands shoulder-width or wider than shoulder-width apart, fingers stretched, palms on the floor, and legs slightly apart. During the test, the participant lowers his torso towards the ground and raises himself up again when his elbows are bent 90º. The movement is repeated as much as possible. The rhythm is set to 20 push-ups per minute or 1 push-up per 3 seconds. The test is terminated when the participant makes a mistake twice. The number of push-ups performed at the end of the test will be recorded. The push-up test will be used to evaluate the upper extremity muscle strength and endurance of children.
FitnessGram Physical Activity Test Battery-Back Saver Sit and Reach Test | Change from baseline and after the exercise program (12 weeks later).
  During the test, the participant takes off his shoes and sits in front of the test apparatus. A box is needed for the test. This box is 35 cm long, 45 cm wide, 32 cm high. A top plate 55 cm long and 45 cm wide is put on top of the box. One leg of the participant is completely straight while the other is bent at the knee. The participant reaches forward four times with their hands on top of each other, holding the fourth reach position for 1 second. At the end of the test, the distance traveled will be recorded. The Back Saver Sit and Reach Test will be used to evaluate the hamstring flexibility of children.
FitnessGram Physical Activity Test Battery-Trunk Lift Test | Change from baseline and after the exercise program (12 weeks later).
  The participant will begin the test in the prone position with their hands placed under the thigh. A sign will be placed on the floor at the participant's eye level. During the movement, the participant will focus on this sign. During the test, the participant slowly and in a controlled manner raises their torso to a maximum height of 12 inches. The head is kept in neutral alignment with the spine. At the end of the test, the distance between the floor and the participant's chin will be measured with a ruler and the score will be recorded in centimeters (cm). Trunk lift test will be used to evaluate trunk extensor muscle strength and flexibility of children.
FitnessGram Physical Activity Test Battery-Progressive Aerobic Cardiovascular Endurance Running (PACER) | Change from baseline and after the exercise program (12 weeks later).
  PACER is an adapted version of the 20 meter shuttle run test and is a field test consisting of multiple stages. The participant will run back and forth in a 20 meter area accompanied by the music coming from the voice recorder. The beep indicates when the participant should finish a lap. The test will start at slow speeds and will gradually increase each minute. The test will be terminated when the participant cannot continue to run at the level he has reached. The number of laps completed at the end of the test will be recorded. PACER is a more fun alternative to other distance running tests. It is recommended for use in children, adolescents and young adults. PACER will be used to assess the aerobic capacity of children.
KFORCE Plates | Change from baseline and after the exercise program (12 weeks later).
  KFORCE Plates is a force platform used to improve balance and evaluate lower extremity muscle symmetry and strength. It consists of two independent plates. KFORCE plates allow measurement of static and dynamic balance in a wide range of movements. It can also determine the center of gravity and measure weight distribution during the stance phase. It evaluates squatting, push-up and jumping characteristics and provides a report containing multiple data as a result of the measurement. Static and dynamic balance analyzes of children will be performed with the device.
KFORCE Muscle Controller | Change from baseline and after the exercise program (12 weeks later).
  KFORCE Muscle Controller is a hand dynamometer used to evaluate muscle strength. It evaluates maximum strength, endurance and muscle symmetry. The muscle controller is versatile and can be adapted to many configurations. As a result of the evaluation, the participant's results are recorded in a database. The participant's progress can then be followed in the application's database. The muscle strength of children will be evaluated with the device.
KBubble | Change from baseline and after the exercise program (12 weeks later).
  The KBubble device is a pressure measurement tool used to assess muscle strength. It evaluates maximum strength, endurance, and muscle symmetry. After the assessment, the participant's results are stored in a database, allowing progress to be monitored over time through the application. In this study, the device will be used to assess lumbar muscle strength in children.
Digitsole Pro® system | Change from baseline and after the exercise program (12 weeks later).
  Digitsole Pro® system consists of wireless sensors, can be fitted in to any shoe and offer the ability to measure spatial, temporal, and kinematic gait parameters. The intelligent insoles feature several sensors that detect and capture foot movements and a micro process or that calculates gait related biomechanical data. Each PODOSmart®insole has an inertial platform that records each foot's walking steps, running strides, and orientations in space with sampling frequency of 208 Hz for walk analysis.The Bluetooth connection box retrieves the collected data by the smart insoles. Then, those data are processed by proprietary artificial intelligence algorithms to calculate the spatiotemporal, kinematic, and biomechanical parameters. Participants' features of walking will be evaluated with the Digitsole Pro® system.
Pain Assessment | Assessed at the end of each of the 24 exercise sessions
  At the end of each exercise session, participants will be asked to rate their pain on a Numerical Rating Scale (NRS) from 0 to 10, where:
  * 0 indicates "no pain at all",
  * 10 indicates "the most severe pain imaginable". This scale helps quantify the intensity of pain experienced after the session.
Fatigue Assessment | Assessed at the end of each of the 24 exercise sessions
  Participants will be asked to rate their level of fatigue on a Numerical Rating Scale (NRS) from 0 to 10, where:
  * 0 indicates "not tired at all",
  * 10 indicates "extremely tired". This provides a subjective measure of how physically exhausting the session was for the participant.
Exercise Satisfaction Rating | Evaluated at the end of the 12-week exercise program.
  Participants will be asked to rate their level of satisfaction with the exercise program using a Numerical Rating Scale (NRS) ranging from 0 to 10 at the end of the 12-week intervention period, where:
  * 0 indicates "not satisfied at all",
  * 10 indicates "extremely satisfied". This provides a subjective measure of how pleased the participant was with the overall exercise experience.

CONTACTS AND LOCATIONS:
Overall Officials: Nilay Arman, Assoc. Prof. Dr., Study Director — Istanbul University-Cerrahpaşa, Faculty of Health Science, Department of Physiotherapy and Rehabilitation, Istanbul, Türkiye; Nuray Aktay Ayaz, Prof. Dr., Study Chair — Istanbul Faculty of Medicine, Department of Internal Medicine, Department of Pediatric Rheumatology, Istanbul, Türkiye.; Figen Cakmak, Assoc. Prof. Dr., Study Chair — Istanbul Basaksehir Cam ve Sakura City Hospital, Department of Pediatric Rheumatology, Istanbul, Türkiye.; Irem Donmez, Pt., Principal Investigator — Istanbul University-Cerrahpasa, Institute of Graduate Studies, Physiotherapy and Rehabilitation Master of Science Program, Istanbul, Türkiye.
Locations (1):
- Istanbul University - Cerrahpasa, Istanbul, Buyukcekmece, Turkey (Türkiye)